CLINICAL TRIAL: NCT01107249
Title: A Phase II Trial of Esophageal and Gastric Stenting for Leak or Perforation
Brief Title: A Trial of Esophageal and Gastric Stenting for Leak or Perforation
Acronym: ESO-stent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00002562; 1108-0322 (Other: HMRI IRB)
Record Dates: First submitted 2010-04-09; First posted 2010-04-20 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Esophageal or Gastric Perforations; Esophageal or Gastric Leaks
Keywords: esophageal; stenting; perforations; gastric; esophageal stenting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BS Ultraflex or Wallstent stents (Other): All subjects receive a stent of surgeons choice from selected stents.
  Interventions: Device: Boston Scientific Ultraflex or Wallstent stents

INTERVENTIONS:
Device: Boston Scientific Ultraflex or Wallstent stents — Stent used to maintain luminal patency in esophageal strictures and occlude esophageal fistulas to reduce gastric leaks, perforations and/or fistulas.
  Other Names: Ultraflex, ULTRAFLEX ESOPHAGEAL NG STENT SYSTEM

SUMMARY:
Long term follow-up of patients treated for esophageal fistulas with a newer occlusive self-expanding covered metal stents compared to traditional stents.

DETAILED DESCRIPTION:
This study is written to evaluate our experience treating esophageal fistulas with occlusive self-expanding covered metal stents. The long-term outcomes of patients treated with this new type of stent are as yet unknown. The differences between these stents is also unknown, as well as the ease of removal, efficacy, and/or placement. The intent of this study is not to determine which stent is better, but to merely evaluate the use of both. With this in mind, there will be no randomization of stent use, nor will there be restrictions on which stent may be used in which setting. This will be left to the judgment of the clinical placing the stent.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have radiographic or endoscopic proof of an esophageal leak or fistula.
2. Patients will be required to undergo imaging with CT scan, endoscopy, or fluoroscopy to investigate the leak. Once the location of the leak is identified, then patients must be taken for stenting and any adjunctive treatment within 12 hours of diagnosis or within 12 hours of arrival to The Methodist Hospital.
3. Patients must sign informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of the hospital.

Exclusion Criteria:

1. Patients who will not agree to return for routine follow-up and studies.
2. Patients who will not tolerate an endobronchial ultrasound or endoscopic procedure (coagulopathy [INR>1.8, PTT>60, or platelet level <50], hemodynamically unstable [MAP<50 or SBP<80], or other medical illness precluding safe endoscopy).
3. Patients who have a perforation too high to stent (such as the back of the pharynx, where a stent is not able to be placed), the only unfavorable anatomic location is this one listed above; we believe all other locations are amenable to stent placement.
4. Resectable carcinoma, megaesophagus, severe stricture, or caustic ingestion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety of esophageal stenting by conducting an Omnipaque swallow and by the success of leakage stops and fistula healing. | 15 - 30 days
  By results from all procedures as reported by the surgeon conducting the stenting in relationship to difficulty and/or complications, as well as patient tolerability. When the esophagus can be sealed and any contamination drained, the stents have successfully provided coverage to allow healing of the esophageal wall.
Efficacy of esophageal stenting by the success of leakage stops and fistula healing. | 15 - 30 days
  By results from all procedures as reported by the surgeon conducting the stenting in relationship to difficulty and/or complications, as well as patient tolerability. When the esophagus can be sealed and any contamination drained, the stents have successfully provided coverage to allow healing of the esophageal wall.
A 30 day duration of stent placement and the relation to the healing esophagus | 30 days
  By results from all procedures as reported by the surgeon conducting the stenting in relationship to difficulty and/or complications, as well as patient tolerability. Evaluation of the healing process of the esophagus within first 30 days with the capability of its removal procedure. When the esophagus can be sealed and any contamination drained, the stents have successfully provided coverage to allow healing of the esophageal wall.

SECONDARY OUTCOMES:
An institutional protocol for stent management | 1 year
  Results will be considered for assessing and instituting an institutional protocol to become the standard of care for future patient situations.

CONTACTS AND LOCATIONS:
Overall Officials: Shanda H Blackmon, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- The Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data at this time. The PI has relocated to another institution and closed the IDE.